CLINICAL TRIAL: NCT02321761
Title: Effect of Amantadine Administration on Spatial Functioning Following Traumatic Brain Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, yaron sacher, The effect of amantadine of spatial attention in patients with traumatic brain injury, Loewenstein Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-12-LOE
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury
Keywords: Amantadine hydrochloride; Rehabilitation; Acquired Brain Injury; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study group (Experimental): Dosage (mg) Day days 0-14 no drug will be given days 15-21 dosage is 100 mg days 22-28 dosage is 200mg days 29-42 dosage is 400mg days 43-56 dosage is 200mg
  days 57-70 no drug will be given
  Interventions: Drug: Amantadine hydrochloride

INTERVENTIONS:
Drug: Amantadine hydrochloride — Drug dosages: day 0-14 no drug will be given Days 15-21 100 mg Days 22-28 200 mg Days 29-42 400 mg Days 43-56 200 day 57-70 no drug will be given
  Other Names: Symmetrel

SUMMARY:
Amantadine hydrochloride is one of the drugs given at rehabilitation programs to people who suffered Acquired Brain Injury in order to expedite recovery and improve functioning.

A previous study examined the spatially asymmetric allocation of attention in patients with traumatic brain injury (TBI). Patients demonstrated significantly worse performance with leftward than with rightward cross-hemi field shifts of attention. This is reminiscence of neglect patients. This difference was significantly reduced during and following treatment. Our objective is to investigate whether Amantadine Hydrochloride is effective in improving allocation of spatial attention and improving function in people with Traumatic Brain Injury.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-50 yrs
2. Patients who were diagnosed with a Diffuse Axonal Injury post TBI
3. Severity of injury was defined as moderate to severe
4. At least 3 months post injury
5. Sufficient cognitive abilities to learn and perform the computerised task.

Exclusion Criteria:

1. Pyramidal signs on neurological examination
2. Localised damage demonstrated on CT
3. Contra indication to Amantadine, post traumatic epilepsy, renal failure and patients with known sensitivity to Amantadine
4. Patients who were diagnosed with Parkinson's disease or has a first degree family who was diagnosed with Parkinson's.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
The Posner Cueing Task | up to day 70
  The study paradigm is based on The Posner Cueing Task, a visual spatial attention task. Identification rates were measured after pre cuing attention to different visual field loci. After pre cuing to a locus 5 degrees into the left or right hemi field, target patterns were presented briefly at the cued location (valid) or on the opposite side (invalid) requiring an attentional shift

CONTACTS AND LOCATIONS:
Locations (1):
- Loewenstein Rehabilitation Center, Raanana, Israel